CLINICAL TRIAL: NCT01936493
Title: Biologic Predictors of Leiomyoma Treatment Outcomes
Status: Completed | Type: Observational
Sponsor: Elizabeth A. Stewart (Other)
Responsible Party: Sponsor-Investigator, Elizabeth A. Stewart, Professor of Obstetrics-Gynecology, Mayo Clinic
Organization: Mayo Clinic (Other)
Other Study IDs: 09-003657
Record Dates: First submitted 2013-08-14; First posted 2013-09-06 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Uterine Leiomyomas; Fibroids; Uterine Fibroids; Myomas
Keywords: Uterine leiomyomas (fibroids or myomas); Uterine fibroids; Fibroids; Uterine leiomyomas
MeSH Terms: conditions — Myofibroma; Leiomyoma; Myoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum aliquots and genomic DNA samples will be collected, processed and stored in the Biospecimen Accessioning Processing (BAP) lab at Mayo Clinic in Rochester, MN.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Females with uterine fibroids: Participants will be females age of 18 or older who have be diagnosed with uterine leiomyoma. Study Subjects will be asked if mothers or siblings also have diagnosis of uterine leoimyoma (either past or present diagnosis) and these family members will be invited to participate in this trial. All participants will provide blood samples for serum aliquots for hormonal analysis and genomic DNA analysis, and will answer a baseline genetic epidemiology questionnaire.
  Interventions: Genetic: DNA analysis; Other: Hormonal analysis

INTERVENTIONS:
Genetic: DNA analysis — At a future time DNA analysis will be performed
Other: Hormonal analysis — Participants will provide blood samples so that hormonal factors that influence outcomes of leiomyoma treatments can be assayed.

SUMMARY:
The purpose of this study is to search for the hereditary (genetic) causes of uterine fibroids. Some women with uterine fibroids may have one or more genes that make them more likely to develop uterine fibroids. We are trying to identify these genes to better understand how and why uterine fibroids develop and to design better treatment options for women with uterine fibroids. This information may also help us to understand and treat other problems that may be caused by these genes.

DETAILED DESCRIPTION:
There is little information to predict outcomes of leiomyoma therapies. It is clear that both environmental exposures and genetic predisposition influence disease manifestations. Our work has identified a new area of genetic linkage for leiomyomas from a genome wide scan. We therefore propose to prospectively collect biologic samples that will allow us to analyze gene/environment interactions of women enrolled in leiomyoma clinical trials or undergoing leiomyoma clinical treatments using the same methodology used previously. Specifically we will collect serum aliquots, genomic DNA and information using a genetic epidemiology questionnaire. In the short term we will also be able to use prospectively obtained information on epidemiologic and anthropomorphic data to characterize women undergoing treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give consent
2. Age 18 or older
3. Presence of known uterine leiomyoma

Exclusion Criteria:

1. Suspected malignancy

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled at Mayo Clinic in Rochester, Minnesota. These patients will either be enrolled in leiomyoma clinical trials or undergoing leiomyoma clinical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2009-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05-26 (Actual)

PRIMARY OUTCOMES:
Analyze environmental exposures and genetic predisposition among women exhibiting disease manifestations of uterine fibroids. | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Stewart, M.D., Principal Investigator — Mayo Clinic - Rochester, Minnesota
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Uterine Fibroids Information — http://www.mayoclinic.com/health/uterine-fibroids/DS00078
- See also: Mayo Clinic Uterine Fibroid Facebook page sharing educational information related to fibroids. — http://on.fb.me/gewuoO